CLINICAL TRIAL: NCT02283385
Title: Mental Health Intervention for Elderly Abuse Victims: Providing Options to Elderly Clients Together (PROTECT)
Brief Title: Mental Health Intervention for Elderly Abuse Victims
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Fan Fox & Leslie R. Samuels Foundation, Inc. (Other); New York City Department for the Aging (Other); Jewish Association Serving the Aging (JASA) (Unknown)
Responsible Party: Principal Investigator, Jo Anne Sirey, Associate Professor, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1306014011
Record Dates: First submitted 2014-10-24; First posted 2014-11-05 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: Elder abuse; Intervention; Treatment; Detection
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROTECT Intervention (Experimental): Participants will receive a brief psychotherapy that builds on Problem Solving Therapy (PST)
  Interventions: Behavioral: PROTECT

INTERVENTIONS:
Behavioral: PROTECT — 8-session weekly psychotherapy intervention that combines problem-solving therapy, anxiety management and psycho education developed specifically for this population

SUMMARY:
There is no current elder abuse service that systematically assesses and provides services to address the mental health needs of older adult abuse victims. The proposed study will investigate the efficacy of a skill-based, mental health intervention to help treat elder abuse victims, bolster mental health outcomes, and improve detection of symptomatology in future screenings.

DETAILED DESCRIPTION:
Despite increasing recognition of the epidemic of elder abuse, we continue to face barriers helping abuse victims access and use elder abuse resolution services. In addition, many victims suffer from concurrent mental health problems that prevent them from taking the necessary steps to protect themselves. The proposed study will introduce a tailored intervention, built on an evidence-based approach (Problem Solving Therapy), to be delivered through a sustainable mental health program embedded in elder abuse services. The proposed psychotherapy is a brief 8-session weekly intervention that combines problem-solving therapy, anxiety management, and psycho education developed specifically for this population by this team.

The objectives of the project are to: identify the mental health needs of elder abuse victims, provide the mental health treatment, assess the impact of the treatment, and facilitate conditions which will sustain the mental health program.

ELIGIBILITY:
Inclusion Criteria:

* Client of the New York City Department for the Aging's (DFTA) Elderly Crime Victims Resource Center
* Score of 10 or higher on the Patient Health Questionnaire (PHQ-9) or Generalized Anxiety Disorder 7-item scale (GAD-7)

Exclusion Criteria:

* Co-morbid psychiatric disorder other than unipolar non-psychotic major depression that prevents participation in depression and anxiety screening
* Inability to speak or understand English
* Cognitive impairment that prevents participation in screening, as determined by screening social worker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Depression (Hamilton Depression Rating Scale) | 12 weeks
  To document effectiveness of PROTECT intervention in reducing depressive symptoms. Severity of depression will be assessed at baseline and 12 weeks using the Hamilton Depression Rating Scale as the primary measure.

SECONDARY OUTCOMES:
Functioning (Behavioral Activation for Depression Scale) | 12 weeks
  To document effectiveness of PROTECT intervention in increasing quality of life, social interaction, and overall functioning. Severity will be assessed at baseline and 12 weeks using the Behavioral Activation for Depression Scale as the primary measure.
Service Utilization (specialized mistreatment and service outcome questionnaires) | 12 weeks
  To document effectiveness of PROTECT intervention in increasing clients' utilization of elder abuse services and subsequently reporting a reduction in abuse. Service utilization and severity of abuse will be assessed at baseline and 12 weeks using specialized mistreatment and service outcome questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Anne Sirey, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Department for the Aging: Elderly Crime Victims Resource Center, New York, New York
  - Jewish Association Serving the Aging, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided